CLINICAL TRIAL: NCT01530971
Title: Effects of Neonate and Maternal Oxygenation in Low-dose Oxygen Supplement by Oxygen Cannula or Non- Supplement in Elective Cesarean Section: a Randomized Controlled Trial
Brief Title: Effect of Maternal and Neonatal Oxygenation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10AS00008/044/10
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Peer Review, Research
Keywords: oxygen; pregnancy; caesarean section; anesthetic techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- room air (No Intervention): no supplemental oxygen in intraoperative period
- Oxygen (Experimental): Supplemental 3LPM oxygen via canula
  Interventions: Drug: Supplemental 3LPM oxygen via canula

INTERVENTIONS:
Drug: Supplemental 3LPM oxygen via canula — Parturients will receive supplemental oxygen (3LPM) via nasal canula
  Arms: Oxygen

SUMMARY:
Intraoperative supplemental oxygen has been given for most parturients undergoing cesarean section under spinal anesthesia. However, evidences supporting the practice is not clear nowadays, especially for healthy parturients who are monitored continuously with pulse oximeter. Furthermore, hyperoxia may produce free radicles which could harm fetus and newborns.

Changing practice is not that easy. This study has been conducted to prove that supplemental oxygen is not necessary for healthy parturients during cesarean section.

DETAILED DESCRIPTION:
Supplemental oxygen has been routinely given to parturients because doctors were concerned about desaturation. However, the evidences for giving oxygen was not strong, and the condition nowadays can be detected immediately with pulse oximeter which is a standard monitoring.

After this study finished, we will set a safety guideline for supplemental oxygen for healthy parturients undergoing elective cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years old.
* Term pregnancy (gestational age 37 -42 weeks).
* Singleton
* Elective cesarean section.

Exclusion Criteria:

* History of infertility
* Diabetes
* Hypertension or preeclampsia
* Heart disease
* Morbid obesity
* Premature rupture of membrane
* Placenta previa
* Preoperative oxygen saturation < 95%

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
proportion of maternal desaturation | intraoperative period
  Oxygen saturation < 94% once.

SECONDARY OUTCOMES:
neonatal outcomes | intraoperative period
  Apgar score and parameters from umbilical cord gas

CONTACTS AND LOCATIONS:
Overall Officials: Arunotai Siriussawakul, MD., Principal Investigator — Mahidol University
Locations (1):
- Siriraj hospital, Bangkok, Thailand

REFERENCES:
- See also: pubmed — http://www.ncbi.nlm.nih.gov/pubmed
- See also: journal @ovid — http://www.ovid.com/site/catalog/journals_landing.jsp
- See also: scopus — http://www.elsevier.com/wps/find/electronicproductdescription.cws_home/704746/description#description